CLINICAL TRIAL: NCT05713071
Title: Evaluation of Bariatric Endoscopic Antral Myotomy (BEAM) as a Treatment for Obesity
Acronym: BEAM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Erbe USA Incorporated (Other)
Responsible Party: Principal Investigator, Christopher C. Thompson, MD, MSc, Director of Endoscopy, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2022P003399
Record Dates: First submitted 2022-12-23; First posted 2023-02-06 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Obesity; Weight Loss; Delayed Gastric Emptying Following Procedure; Obesity, Mild; Obesity, Morbid; Obesity; Excess Calories
Keywords: Bariatric Endoscopic Antral Myotomy (BEAM); Gastric physiology; Gastric emptying; Pylorus-sparing antral myotomy; Myotomy; Endoscopic Sleeve Gastroplasty (ESG); TransPyloric Shuttle (TPS); Intragastric balloon (IGB); Endoscopic bariatric and metabolic therapies (EBMT); Gut Hormones; Gastric Emptying Breath Test
MeSH Terms: conditions — Obesity; Weight Loss; Lymphoma, Follicular; Obesity, Morbid

STUDY DESIGN:
Intervention Model Description: This pilot, single-center, randomized, controlled, clinical study aims to assess the safety, tolerability, and short-term efficacy of BEAM, in addition to exploring its impact on gastric physiology compared to lifestyle modification therapy alone. At 6 months control group will crossover to treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BEAM Treatment Patients (Experimental): Subjects having esophagogastroduodenoscopy (EGD) with Bariatric Endoscopic Antral Myotomy (BEAM) with standard of care lifestyle modification therapy.
  Interventions: Procedure: Bariatric Endoscopic Antral Myotomy
- Lifestyle Modification Control Group (No Intervention): Standard of care lifestyle modification therapy only.

INTERVENTIONS:
Procedure: Bariatric Endoscopic Antral Myotomy — BEAM will be performed using a standard gastric peroral endoscopic myotomy (G-POEM) technique, however with the myotomy targeting only the antrum and leaving the pyloric ring intact. G-POEM is commonly and widely employed for gastric emptying and nutritional issues and is covered by most insurance plans. This involves injecting fluid into the submucosal space, making a mucosal incision to enter the submucosal space, and tunneling along the antrum to the pylorus. A myotomy is then performed, however, in BEAM the pyloric ring is spared and the myotomy is only performed in the antrum. The incision is then closed with clips. No endoscopic suturing will be performed.
  Other Names: BEAM
  Arms: BEAM Treatment Patients

SUMMARY:
In the proposed study, we will be evaluating the effects of pylorus sparing antral myotomy alone, without concomitant endoscopic sleeve gastroplasty (ESG), on weight loss for subjects undergoing the procedure with a history of obesity. This is referred to as Bariatric Endoscopic Antral Myotomy (BEAM). To better understand treatment effects, we will track weight loss, gastric emptying with gastric emptying breath tests (GEBT), and gut hormones (i.e. ghrelin).

This pilot, single-center, randomized, controlled, clinical study aims to assess the safety, tolerability, and short-term efficacy of BEAM, in addition to exploring its impact on gastric physiology. This will also provide data that may be used in designing a larger clinical trial that could be submitted for NIH grant funding.

DETAILED DESCRIPTION:
Obesity is generally defined as a body mass index (BMI) of at least 30 kg/m2. It affects 30% of the global population and poses a significant healthcare burden. [1] Obesity has increased dramatically over the last few decades with over 650 million adults, or 13% of the world's total adult population, meeting diagnostic criteria in 2016.[1] In the U.S. the prevalence of obesity increased by 89.9% between 1993 and 2008.[1,2,3] As a result, current and potential interventions, and treatment strategies to combat obesity have become more important.

Sleeve gastrectomy, a bariatric surgical procedure, involves resection of the greater curvature of the stomach resulting in more rapid gastric emptying. It has been thought to reduce weight loss by increasing satiation as well as by triggering hindgut mechanisms. These mechanisms include increase in production of certain gut hormones, including GLP-1.[4] Sleeve gastrectomy and other bariatric surgeries are very effective at treating obesity, however, only 1% of eligible subjects elect to undergo this treatment option. Additionally, most subjects with obesity do not qualify for bariatric surgery.[5]

Endoscopic bariatric and metabolic therapies (EBMT) have recently emerged as alternative treatments for patients with obesity and a BMI over 30kg/m2. Interest in EBMT is growing given their safety, efficacy, and non-invasive nature. Current FDA- approved devices include intragastric balloons (IGB) and suturing devices for endoscopic sleeve gastroplasty (ESG). These gastric interventions work by interfering with gastric accommodation, breakdown and mixing of food, or the antral pump. All of which ultimately impact gastric emptying. IGB are space occupying devices that cause early satiation and must be removed after approximately six months, with subsequent weight regain being an issue. ESG involves endoscopic suturing to reduce the length and width of the stomach to similarly trigger earlier satiation. Delay of gastric emptying has been shown to be a major mechanism of action for both ESG and IGB, and this is also correlated with weight loss, although it is less consistent and well characterized following ESG. [6]

ESG is associated with approximately 16% TWL at one year and is well tolerated with a 1-2% SAE rate.[7] However, there are several limitations to the procedure in its current form. It is technically demanding with a long learning curve of approximately 50 cases, resulting in few centers offering the procedure, and suture loss is common raising questions of long-term durability.[8] There are also numerous suture patterns employed in clinical practice impacting the consistency of results and available suturing platforms are expensive limiting health equity.

The TransPyloric Shuttle (TPS) is a specialized balloon that resides in the gastric antrum and is the only device that incapacitates the antral pump directly impacting gastric emptying. As with other IGB, the TPS must be removed after several months resulting in subsequent weight regain.[9]

Gastroplasty with Endoscopic Myotomy (GEM) involves an abbreviated ESG of the gastric body with a pylorus-sparing antral myotomy, adding the TPS mechanism to that of traditional ESG. This employs a modification of the Gastric Peroral Endoscopic Myotomy (G-POEM) technique, targeting the antrum and leaving the pyloric ring intact to slow emptying, instead of making it more rapid. The goal of this procedure is to address the major limitations of ESG, including the procedural variability, technical difficulty, and durability. A small study has shown a consistent delay in gastric emptying with GEM, with the T ½ going from approximately 90 minutes to over 200 minutes, with 20% TWL that continues to trend downward at 6 months. Additionally, there were no new symptoms detected on the Gastroparesis Cardinal Symptom Index (GCSI) score following the procedure.

Although early results suggest the addition of antral myotomy to ESG in the GEM procedure appears to increase weight loss and consistency of delayed gastric emptying, there have been no clinical studies that investigate the efficacy of pylorus sparing antral myotomy alone, without concomitant ESG. However, this approach could have many benefits due to its less invasive nature and relative technical simplicity. There are more endoscopists with the skillset necessary to perform antral myotomy than can perform ESG, and the learning curve would also be substantially shorter. Additionally, the cost of this approach would be considerably lower than current therapies as it only involves an endoscopic procedure, an electrosurgical knife and clips for closure, with no need for an expensive suturing system.

In the proposed study, we will be evaluating the effects of pylorus sparing antral myotomy alone, without concomitant ESG, on weight loss for subjects undergoing the procedure with a history of obesity. This is referred to as Bariatric Endoscopic Antral Myotomy (BEAM). To better understand treatment effects, we will track weight loss, gastric emptying with gastric emptying breath tests (GEBT), and gut hormones (i.e. ghrelin).

This pilot, single-center, randomized, controlled, clinical study aims to assess the safety, tolerability, and short-term efficacy of BEAM, in addition to exploring its impact on gastric physiology. This will also provide data that may be used in designing a larger clinical trial that could be submitted for NIH grant funding.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be 18-70 years of age
2. Are currently in the CWMW lifestyle modification program
3. Have a diagnostic endoscopy approved for bariatric evaluation
4. Eligible for endoscopic and surgical weight loss procedures
5. Body mass index (BMI) 30-50 kg/m2
6. Individuals must be in excellent mental health
7. Able to understand and sign informed consent
8. Available to return for all routine follow-up study visits

Exclusion Criteria:

1. Untreated H. pylori infection
2. Active smoking
3. Ongoing or a history of treatment with opioids in the last 12 months prior to enrollment
4. Previous pyloromyotomy or pyloroplasty
5. Gastrointestinal obstruction
6. Severe coagulopathy
7. Esophageal or gastric varices and/or portal hypertensive gastropathy
8. Pregnancy or puerperium
9. Any inflammatory disease of the gastrointestinal tract (including but not limited to severe (LA Grade C or D) esophagitis, active gastric ulceration, active duodenal ulceration, or specific inflammation such as Crohn's disease)
10. Malignant or premalignant gastric diseases (such as high grade dysplasia, gastric cancer, or GIST)
11. Severe cardiopulmonary disease or a history of coronary artery disease (including myocardial infarction within the past 6 months, poorly controlled hypertension, required use of NSAIDs)
12. Lactation
13. History of gastrointestinal surgery
14. Any serious health condition unrelated to their weight that would increase the risk of endoscopy
15. Chronic abdominal pain
16. Active psychological issues preventing participation in a lifestyle modification program
17. A known history of endocrine disorders affecting weight (uncontrolled hypothyroidism)
18. An inability to provide informed consent
19. Use of any medication that may interfere with weight loss
20. Use of any medication that may interfere with gastric emptying
21. Any other condition which the investigator may deem as an impediment to compliance or hinder completion of the proposed study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-02-21 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Weight change compared to baseline | Screening, Day 0/Treatment, 1 month, 3 month, 6 month, 9 month, 12 months
  percent total body weight loss
Adverse Events | Day 0/Treatment, 1 month, 3 month, 6 month, 9 month, 12 months
  Changes to health compared to baseline
Changed in pain scale from Day 0 to 12 months | Day 0/Treatment, 1 month, 3 month, 6 month, 9 month, 12 months
  How the subjects feel after the procedure based on pain scale (no pain = 1- worst possible pain = 10)

SECONDARY OUTCOMES:
Change in Quality of Life compared to baseline using the Impact of Weight on Quality of Life Lite (IWQOL-Lite) Questionnaire | Screening, 1 month, 3 month, 6 month, 9 month, 12 months
  Overall quality of life questionnaire (IWQOL-Lite) - scale 1 (Never True) - 5 (Always True)
Gastric Emptying compared to baseline | Screening, 6 months, 12 months
  Gastric emptying using a gastric emptying breath test (GEBT)
Ghrelin levels compared to baseline | Screening, 6 months, 12 months
  Laboratory analysis of blood samples to test ghrelin levels
Change in insulin metabolic profiles compared to baseline | Screening, 6 months, 12 months
  Laboratory analysis of insulin blood samples to test metabolic profiles
Change in HgA1c levels compared to baseline | Screening, 6 months, 12 months
  Laboratory analysis of HgA1c blood samples to test metabolic profiles
Change in glucose levels compared to baseline | Screening, 6 months, 12 months
  Laboratory analysis of glucose blood samples to test metabolic profiles
Change in HOMA-IR levels compared to baseline | Screening, 6 months, 12 months
  Laboratory analysis of HOMA-IR blood samples to test insulin resistance
Radiological (Upper GI Series) gastric emptying rate (minutes) of barium transit from esophagus through stomach to small intestine compared to baseline | Screening, 6 months, 12 months
  Upper GI series comparing barium transit from baseline to 6 and 12 months post-procedure.
Radiological (Dynamic MRI) gastric emptying rate (minutes) of contrast transit from esophagus, through stomach to small intestine compared to baseline compared to baseline | Screening, 1 month
  Dynamic MRI comparing contrast transit from baseline to 1 month post-procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher C. Thompson, MD, MSc, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
As this is a pilot study for potential NIH Grant submission, we do not plan to share data with other researchers at this time.

REFERENCES:
- [Background] Klem ML, Wing RR, Chang CC, Lang W, McGuire MT, Sugerman HJ, Hutchison SL, Makovich AL, Hill JO. A case-control study of successful maintenance of a substantial weight loss: individuals who lost weight through surgery versus those who lost weight through non-surgical means. Int J Obes Relat Metab Disord. 2000 May;24(5):573-9. doi: 10.1038/sj.ijo.0801199. PMID 10849578
- [Background] James PT, Leach R, Kalamara E, Shayeghi M. The worldwide obesity epidemic. Obes Res. 2001 Nov;9 Suppl 4:228S-233S. doi: 10.1038/oby.2001.123. PMID 11707546
- [Background] Jia H, Lubetkin EI. Obesity-related quality-adjusted life years lost in the U.S. from 1993 to 2008. Am J Prev Med. 2010 Sep;39(3):220-7. doi: 10.1016/j.amepre.2010.03.026. PMID 20709253
- [Background] McCarty TR, Jirapinyo P, Thompson CC. Effect of Sleeve Gastrectomy on Ghrelin, GLP-1, PYY, and GIP Gut Hormones: A Systematic Review and Meta-analysis. Ann Surg. 2020 Jul;272(1):72-80. doi: 10.1097/SLA.0000000000003614. PMID 31592891
- [Background] Abu Dayyeh BK, Rajan E, Gostout CJ. Endoscopic sleeve gastroplasty: a potential endoscopic alternative to surgical sleeve gastrectomy for treatment of obesity. Gastrointest Endosc. 2013 Sep;78(3):530-5. doi: 10.1016/j.gie.2013.04.197. Epub 2013 May 24. PMID 23711556
- [Background] Gomez V, Woodman G, Abu Dayyeh BK. Delayed gastric emptying as a proposed mechanism of action during intragastric balloon therapy: Results of a prospective study. Obesity (Silver Spring). 2016 Sep;24(9):1849-53. doi: 10.1002/oby.21555. Epub 2016 Jul 28. PMID 27465076
- [Background] Hedjoudje A, Abu Dayyeh BK, Cheskin LJ, Adam A, Neto MG, Badurdeen D, Morales JG, Sartoretto A, Nava GL, Vargas E, Sui Z, Fayad L, Farha J, Khashab MA, Kalloo AN, Alqahtani AR, Thompson CC, Kumbhari V. Efficacy and Safety of Endoscopic Sleeve Gastroplasty: A Systematic Review and Meta-Analysis. Clin Gastroenterol Hepatol. 2020 May;18(5):1043-1053.e4. doi: 10.1016/j.cgh.2019.08.022. Epub 2019 Aug 20. PMID 31442601
- [Background] Saumoy M, Schneider Y, Zhou XK, Shukla A, Kahaleh M, Aronne L, Sharaiha RZ. A single-operator learning curve analysis for the endoscopic sleeve gastroplasty. Gastrointest Endosc. 2018 Feb;87(2):442-447. doi: 10.1016/j.gie.2017.08.014. Epub 2017 Aug 24. PMID 28843586
- [Background] Marinos G, Eliades C, Raman Muthusamy V, Greenway F. Weight loss and improved quality of life with a nonsurgical endoscopic treatment for obesity: clinical results from a 3- and 6-month study. Surg Obes Relat Dis. 2014 Sep-Oct;10(5):929-34. doi: 10.1016/j.soard.2014.03.005. Epub 2014 Mar 12. PMID 25066439
- [Background] Aghaie Meybodi M, Qumseya BJ, Shakoor D, Lobner K, Vosoughi K, Ichkhanian Y, Khashab MA. Efficacy and feasibility of G-POEM in management of patients with refractory gastroparesis: a systematic review and meta-analysis. Endosc Int Open. 2019 Mar;7(3):E322-E329. doi: 10.1055/a-0812-1458. Epub 2019 Feb 28. PMID 30842971
- [Background] Mohan BP, Chandan S, Jha LK, Khan SR, Kotagiri R, Kassab LL, Ravikumar NPG, Bhogal N, Chandan OC, Bhat I, Hewlett AT, Jacques J, Ponnada S, Asokkumar R, Adler DG. Clinical efficacy of gastric per-oral endoscopic myotomy (G-POEM) in the treatment of refractory gastroparesis and predictors of outcomes: a systematic review and meta-analysis using surgical pyloroplasty as a comparator group. Surg Endosc. 2020 Aug;34(8):3352-3367. doi: 10.1007/s00464-019-07135-9. Epub 2019 Oct 3. PMID 31583465